CLINICAL TRIAL: NCT00802178
Title: CEE PMSS (Central Eastern European Post-Marketing Surveillance Study) First Presentation of Mirapexin in Parkinson Patients
Brief Title: First Presentation of Parkinson Disease Patients to Neurologist
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.613
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Results first posted 2009-11-20 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In this study information is gathered about the treatment of Parkinson patients who present themselves in a neurological practice for the first time

ELIGIBILITY:
Inclusion Criteria:

- Parkinson Disease patients presenting to neurologist for first time

Exclusion Criteria:

- Hypersensitivity to the active substance or to any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neurogologists
Sampling Method: Non-Probability Sample
Enrollment: 2448 (Actual)
Dates: Start 2006-02; Primary Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (311):
- Croatia (11):
  - Boehringer Ingelheim Investigational Site, Bjelovar
  - Boehringer Ingelheim Investigational Site, Dubrovnik
  - Boehringer Ingelheim Investigational Site, Gospić
  - Boehringer Ingelheim Investigational Site, Karlovac
  - Boehringer Ingelheim Investigational Site, Požega
  - Boehringer Ingelheim Investigational Site, Pula
  - Boehringer Ingelheim Investigational Site, Rijeka
  - Boehringer Ingelheim Investigational Site, Sisak
  - Boehringer Ingelheim Investigational Site, Split
  - Boehringer Ingelheim Investigational Site, Šibenik
  - Boehringer Ingelheim Investigational Site, Zabok
- Czechia (104):
  - Boehringer Ingelheim Investigational Site, Blansko
  - Boehringer Ingelheim Investigational Site, Brandýs N. Orlicí
  - Boehringer Ingelheim Investigational Site 1, Brno
  - Boehringer Ingelheim Investigational Site 2, Brno
  - Boehringer Ingelheim Investigational Site, Bystřice N. Pernštejnem
  - Boehringer Ingelheim Investigational Site 1, Cheb
  - Boehringer Ingelheim Investigational Site 2, Cheb
  - Boehringer Ingelheim Investigational Site 3, Cheb
  - Boehringer Ingelheim Investigational Site 1, Chomutov
  - Boehringer Ingelheim Investigational Site 2, Chomutov
  - Boehringer Ingelheim Investigational Site, Černožice
  - Boehringer Ingelheim Investigational Site 1, Česká Lípa
  - Boehringer Ingelheim Investigational Site 2, Česká Lípa
  - Boehringer Ingelheim Investigational Site 1, České Budějovice
  - Boehringer Ingelheim Investigational Site 2, České Budějovice
  - Boehringer Ingelheim Investigational Site 3, České Budějovice
  - Boehringer Ingelheim Investigational Site 4, České Budějovice
  - Boehringer Ingelheim Investigational Site, Český Krumlov
  - Boehringer Ingelheim Investigational Site, Frýdek-Místek
  - Boehringer Ingelheim Investigational Site, Havíov
  - Boehringer Ingelheim Investigational Site, Hodonín
  - Boehringer Ingelheim Investigational Site, Holešov
  - Boehringer Ingelheim Investigational Site, Hradec Králové
  - Boehringer Ingelheim Investigational Site, Jablonec N. Nisou
  - Boehringer Ingelheim Investigational Site, Jičín
  - Boehringer Ingelheim Investigational Site, Jilemnice
  - Boehringer Ingelheim Investigational Site 1, Karlovy Vary
  - Boehringer Ingelheim Investigational Site 2, Karlovy Vary
  - Boehringer Ingelheim Investigational Site, Kladno
  - Boehringer Ingelheim Investigational Site, Kolín
  - Boehringer Ingelheim Investigational Site 1, Kroměříz
  - Boehringer Ingelheim Investigational Site 2, Kroměříz
  - Boehringer Ingelheim Investigational Site 1, Kyjov
  - Boehringer Ingelheim Investigational Site 2, Kyjov
  - Boehringer Ingelheim Investigational Site 1, Liberec
  - Boehringer Ingelheim Investigational Site 2, Liberec
  - Boehringer Ingelheim Investigational Site 3, Liberec
  - Boehringer Ingelheim Investigational Site, Lipník nad Bečvou
  - Boehringer Ingelheim Investigational Site 1, Litoměřice
  - Boehringer Ingelheim Investigational Site 2, Litoměřice
  - Boehringer Ingelheim Investigational Site 1, Litomyšl
  - Boehringer Ingelheim Investigational Site 2, Litomyšl
  - Boehringer Ingelheim Investigational Site, Litovel
  - Boehringer Ingelheim Investigational Site, Mladá Boleslav
  - Boehringer Ingelheim Investigational Site, Moravské Budějovice
  - Boehringer Ingelheim Investigational Site, Moravský Krumlov
  - Boehringer Ingelheim Investigational Site, Náchod
  - Boehringer Ingelheim Investigational Site 1, Olomouc
  - Boehringer Ingelheim Investigational Site 2, Olomouc
  - Boehringer Ingelheim Investigational Site 3, Olomouc
  - Boehringer Ingelheim Investigational Site 4, Olomouc
  - Boehringer Ingelheim Investigational Site 5, Olomouc
  - Boehringer Ingelheim Investigational Site 6, Olomouc
  - Boehringer Ingelheim Investigational Site 7, Olomouc
  - Boehringer Ingelheim Investigational Site, Opava
  - Boehringer Ingelheim Investigational Site, Ostrava - Poruba
  - Boehringer Ingelheim Investigational Site, Ostrava Pustkovec
  - Boehringer Ingelheim Investigational Site 1, Pilsen
  - Boehringer Ingelheim Investigational Site 2, Pilsen
  - Boehringer Ingelheim Investigational Site 3, Pilsen
  - Boehringer Ingelheim Investigational Site 4, Pilsen
  - Boehringer Ingelheim Investigational Site 5, Pilsen
  - Boehringer Ingelheim Investigational Site 6, Pilsen
  - Boehringer Ingelheim Investigational Site 7, Pilsen
  - Boehringer Ingelheim Investigational Site, Písek
  - Boehringer Ingelheim Investigational Site 10, Prague
  - Boehringer Ingelheim Investigational Site 11, Prague
  - Boehringer Ingelheim Investigational Site 13, Prague
  - Boehringer Ingelheim Investigational Site 14, Prague
  - Boehringer Ingelheim Investigational Site 15, Prague
  - Boehringer Ingelheim Investigational Site 16, Prague
  - Boehringer Ingelheim Investigational Site 17, Prague
  - Boehringer Ingelheim Investigational Site 18, Prague
  - Boehringer Ingelheim Investigational Site 19, Prague
  - Boehringer Ingelheim Investigational Site 1, Prague
  - Boehringer Ingelheim Investigational Site 20, Prague
  - Boehringer Ingelheim Investigational Site 21, Prague
  - Boehringer Ingelheim Investigational Site 2, Prague
  - Boehringer Ingelheim Investigational Site 3, Prague
  - Boehringer Ingelheim Investigational Site 4, Prague
  - Boehringer Ingelheim Investigational Site 5, Prague
  - Boehringer Ingelheim Investigational Site 6, Prague
  - Boehringer Ingelheim Investigational Site 7, Prague
  - Boehringer Ingelheim Investigational Site 8, Prague
  - Boehringer Ingelheim Investigational Site 9, Prague
  - Boehringer Ingelheim Investigational Site 12, Praha 4 - Kamýk
  - Boehringer Ingelheim Investigational Site, Přerov
  - Boehringer Ingelheim Investigational Site, Přeštice
  - Boehringer Ingelheim Investigational Site 1, Příbram
  - Boehringer Ingelheim Investigational Site 2, Příbram
  - Boehringer Ingelheim Investigational Site, Srubec, České Budějovice
  - Boehringer Ingelheim Investigational Site, Stenberk
  - Boehringer Ingelheim Investigational Site, Strakonice
  - Boehringer Ingelheim Investigational Site, Svitavy
  - Boehringer Ingelheim Investigational Site, Teplice
  - Boehringer Ingelheim Investigational Site, Trutnov
  - Boehringer Ingelheim Investigational Site, Třebíč
  - Boehringer Ingelheim Investigational Site, Třinec
  - Boehringer Ingelheim Investigational Site, Ústí N. Labem
  - Boehringer Ingelheim Investigational Site, Vojnův Městec
  - Boehringer Ingelheim Investigational Site, Zlín
  - Boehringer Ingelheim Investigational Site, Znojmo
  - Boehringer Ingelheim Investigational Site 1, Žďár N. Sázavou
  - Boehringer Ingelheim Investigational Site 2, Žďár N. Sázavou
- Estonia (4):
  - Boehringer Ingelheim Investigational Site, Kohtla-Järve
  - Boehringer Ingelheim Investigational Site, Pärnu
  - Boehringer Ingelheim Investigational Site, Tallinn
  - Boehringer Ingelheim Investigational Site, Tartu
- Hungary (40):
  - Boehringer Ingelheim Investigational Site, Balassagyarmat
  - Boehringer Ingelheim Investigational Site, Berettyóújfalu
  - Boehringer Ingelheim Investigational Site 10, Budapest
  - Boehringer Ingelheim Investigational Site 11, Budapest
  - Boehringer Ingelheim Investigational Site 12, Budapest
  - Boehringer Ingelheim Investigational Site 13, Budapest
  - Boehringer Ingelheim Investigational Site 14, Budapest
  - Boehringer Ingelheim Investigational Site 15, Budapest
  - Boehringer Ingelheim Investigational Site 1, Budapest
  - Boehringer Ingelheim Investigational Site 2, Budapest
  - Boehringer Ingelheim Investigational Site 3, Budapest
  - Boehringer Ingelheim Investigational Site 4, Budapest
  - Boehringer Ingelheim Investigational Site 5, Budapest
  - Boehringer Ingelheim Investigational Site 6, Budapest
  - Boehringer Ingelheim Investigational Site 7, Budapest
  - Boehringer Ingelheim Investigational Site 8, Budapest
  - Boehringer Ingelheim Investigational Site 9, Budapest
  - Boehringer Ingelheim Investigational Site 1, Debrecen
  - Boehringer Ingelheim Investigational Site 2, Debrecen
  - Boehringer Ingelheim Investigational Site, Dunaújváros
  - Boehringer Ingelheim Investigational Site, Eger
  - Boehringer Ingelheim Investigational Site, Esztergom
  - Boehringer Ingelheim Investigational Site, Gyõr
  - Boehringer Ingelheim Investigational Site, Hatvan
  - Boehringer Ingelheim Investigational Site, Kaposvár
  - Boehringer Ingelheim Investigational Site 1, Kecskemét
  - Boehringer Ingelheim Investigational Site 2, Kecskemét
  - Boehringer Ingelheim Investigational Site, Kistarcsa
  - Boehringer Ingelheim Investigational Site, Kisvárda
  - Boehringer Ingelheim Investigational Site, Miskolc
  - Boehringer Ingelheim Investigational Site, Nyíregyháza
  - Boehringer Ingelheim Investigational Site 1, Pécs
  - Boehringer Ingelheim Investigational Site 2, Pécs
  - Boehringer Ingelheim Investigational Site, Ráckeve
  - Boehringer Ingelheim Investigational Site, Salgótarján
  - Boehringer Ingelheim Investigational Site, Sopron
  - Boehringer Ingelheim Investigational Site, Szekszárd
  - Boehringer Ingelheim Investigational Site, Szentendre
  - Boehringer Ingelheim Investigational Site, Vác
  - Boehringer Ingelheim Investigational Site, Veszprém
- Romania (75):
  - Boehringer Ingelheim Investigational Site, Alba Iulia
  - Boehringer Ingelheim Investigational Site, Arad
  - Boehringer Ingelheim Investigational Site, Bacau
  - Boehringer Ingelheim Investigational Site 1, Baia Mare
  - Boehringer Ingelheim Investigational Site 2, Baia Mare
  - Boehringer Ingelheim Investigational Site, Bistriţa
  - Boehringer Ingelheim Investigational Site, Brasov
  - Boehringer Ingelheim Investigational Site 10, Bucharest
  - Boehringer Ingelheim Investigational Site 11, Bucharest
  - Boehringer Ingelheim Investigational Site 12, Bucharest
  - Boehringer Ingelheim Investigational Site 13, Bucharest
  - Boehringer Ingelheim Investigational Site 14, Bucharest
  - Boehringer Ingelheim Investigational Site 15, Bucharest
  - Boehringer Ingelheim Investigational Site 16, Bucharest
  - Boehringer Ingelheim Investigational Site 17, Bucharest
  - Boehringer Ingelheim Investigational Site 18, Bucharest
  - Boehringer Ingelheim Investigational Site 19, Bucharest
  - Boehringer Ingelheim Investigational Site 1, Bucharest
  - Boehringer Ingelheim Investigational Site 20, Bucharest
  - Boehringer Ingelheim Investigational Site 21, Bucharest
  - Boehringer Ingelheim Investigational Site 2, Bucharest
  - Boehringer Ingelheim Investigational Site 3, Bucharest
  - Boehringer Ingelheim Investigational Site 4, Bucharest
  - Boehringer Ingelheim Investigational Site 5, Bucharest
  - Boehringer Ingelheim Investigational Site 6, Bucharest
  - Boehringer Ingelheim Investigational Site 7, Bucharest
  - Boehringer Ingelheim Investigational Site 8, Bucharest
  - Boehringer Ingelheim Investigational Site 9, Bucharest
  - Boehringer Ingelheim Investigational Site 1, Buzău
  - Boehringer Ingelheim Investigational Site 2, Buzău
  - Boehringer Ingelheim Investigational Site 3, Buzău
  - Boehringer Ingelheim Investigational Site, Campulung Muscel
  - Boehringer Ingelheim Investigational Site, Câmpina
  - Boehringer Ingelheim Investigational Site 1, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 2, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 3, Cluj-Napoca
  - Boehringer Ingelheim Investigational Site 1, Constanța
  - Boehringer Ingelheim Investigational Site 2, Constanța
  - Boehringer Ingelheim Investigational Site 3, Constanța
  - Boehringer Ingelheim Investigational Site 1, Craiova
  - Boehringer Ingelheim Investigational Site 2, Craiova
  - Boehringer Ingelheim Investigational Site 3, Craiova
  - Boehringer Ingelheim Investigational Site 1, Curtea de Argeş
  - Boehringer Ingelheim Investigational Site 2, Curtea de Argeş
  - Boehringer Ingelheim Investigational Site, Deva
  - Boehringer Ingelheim Investigational Site, Drobeta-Turnu Severin
  - Boehringer Ingelheim Investigational Site 1, Galati
  - Boehringer Ingelheim Investigational Site 2, Galati
  - Boehringer Ingelheim Investigational Site, Giurgiu
  - Boehringer Ingelheim Investigational Site 1, Iași
  - Boehringer Ingelheim Investigational Site 2, Iași
  - Boehringer Ingelheim Investigational Site 3, Iași
  - Boehringer Ingelheim Investigational Site 4, Iași
  - Boehringer Ingelheim Investigational Site 1, Oradea
  - Boehringer Ingelheim Investigational Site 2, Oradea
  - Boehringer Ingelheim Investigational Site, Petroşani
  - Boehringer Ingelheim Investigational Site, Piatra Neamţ
  - Boehringer Ingelheim Investigational Site 1, Piteşti
  - Boehringer Ingelheim Investigational Site 2, Piteşti
  - Boehringer Ingelheim Investigational Site 1, Ploieşti
  - Boehringer Ingelheim Investigational Site 2, Ploieşti
  - Boehringer Ingelheim Investigational Site 3, Ploieşti
  - Boehringer Ingelheim Investigational Site, Rm Valcea
  - Boehringer Ingelheim Investigational Site 1, Satu Mare
  - Boehringer Ingelheim Investigational Site 2, Satu Mare
  - Boehringer Ingelheim Investigational Site, Sibiu
  - Boehringer Ingelheim Investigational Site, Slatina
  - Boehringer Ingelheim Investigational Site, Slobozia
  - Boehringer Ingelheim Investigational Site, Suceava
  - Boehringer Ingelheim Investigational Site, Tg Mures
  - Boehringer Ingelheim Investigational Site 1, Timișoara
  - Boehringer Ingelheim Investigational Site 2, Timișoara
  - Boehringer Ingelheim Investigational Site 3, Timișoara
  - Boehringer Ingelheim Investigational Site 4, Timișoara
  - Boehringer Ingelheim Investigational Site 5, Timișoara
- Russia (4):
  - Boehringer Ingelheim Investigational Site 1, Moscow
  - Boehringer Ingelheim Investigational Site 2, Moscow
  - Boehringer Ingelheim Investigational Site 1, Saint Petersburg
  - Boehringer Ingelheim Investigational Site 2, Saint Petersburg
- Serbia (18):
  - Boehringer Ingelheim Investigational Site, Arandjelovac
  - Boehringer Ingelheim Investigational Site 1, Belgrade
  - Boehringer Ingelheim Investigational Site 2, Belgrade
  - Boehringer Ingelheim Investigational Site 3, Belgrade
  - Boehringer Ingelheim Investigational Site 4, Belgrade
  - Boehringer Ingelheim Investigational Site, Kikinda
  - Boehringer Ingelheim Investigational Site, Knjazevac
  - Boehringer Ingelheim Investigational Site, Kragujevac
  - Boehringer Ingelheim Investigational Site, Kruševac
  - Boehringer Ingelheim Investigational Site, Loznica
  - Boehringer Ingelheim Investigational Site, Negotin
  - Boehringer Ingelheim Investigational Site, Niš
  - Boehringer Ingelheim Investigational Site, Novi Sad
  - Boehringer Ingelheim Investigational Site, Sombor
  - Boehringer Ingelheim Investigational Site, Sremska Mitrovica
  - Boehringer Ingelheim Investigational Site, Subotica
  - Boehringer Ingelheim Investigational Site, Vranje
  - Boehringer Ingelheim Investigational Site, Zaječar
- Slovakia (45):
  - Boehringer Ingelheim Investigational Site 1, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 2, Banská Bystrica
  - Boehringer Ingelheim Investigational Site 3, Banská Bystrica
  - Boehringer Ingelheim Investigational Site, Bánovce N. Bebravou
  - Boehringer Ingelheim Investigational Site 1, Bratislava
  - Boehringer Ingelheim Investigational Site 2, Bratislava
  - Boehringer Ingelheim Investigational Site 3, Bratislava
  - Boehringer Ingelheim Investigational Site 4, Bratislava
  - Boehringer Ingelheim Investigational Site 5, Bratislava
  - Boehringer Ingelheim Investigational Site, Dolný Kubín
  - Boehringer Ingelheim Investigational Site, Galanta
  - Boehringer Ingelheim Investigational Site, Komárno
  - Boehringer Ingelheim Investigational Site 5, Kosice- Saca
  - Boehringer Ingelheim Investigational Site 1, Košice
  - Boehringer Ingelheim Investigational Site 2, Košice
  - Boehringer Ingelheim Investigational Site 3, Košice
  - Boehringer Ingelheim Investigational Site 4, Košice
  - Boehringer Ingelheim Investigational Site, Levice
  - Boehringer Ingelheim Investigational Site, Liptovský Mikulás
  - Boehringer Ingelheim Investigational Site, Martin
  - Boehringer Ingelheim Investigational Site, Myjava
  - Boehringer Ingelheim Investigational Site 1, Nitra
  - Boehringer Ingelheim Investigational Site 2, Nitra
  - Boehringer Ingelheim Investigational Site, Nováky
  - Boehringer Ingelheim Investigational Site, Povazská Bystrica
  - Boehringer Ingelheim Investigational Site 1, Prešov
  - Boehringer Ingelheim Investigational Site 2, Prešov
  - Boehringer Ingelheim Investigational Site, Prievidza
  - Boehringer Ingelheim Investigational Site, Rimavská Sobota
  - Boehringer Ingelheim Investigational Site, Roz?ava
  - Boehringer Ingelheim Investigational Site, Ružomberok
  - Boehringer Ingelheim Investigational Site, Skalica
  - Boehringer Ingelheim Investigational Site, Sliač
  - Boehringer Ingelheim Investigational Site, Snina
  - Boehringer Ingelheim Investigational Site 2, Stará ?ubov?a
  - Boehringer Ingelheim Investigational Site 1, Stará Ľubovňa
  - Boehringer Ingelheim Investigational Site, Šurany
  - Boehringer Ingelheim Investigational Site, Topoľčany
  - Boehringer Ingelheim Investigational Site 1, Trebišov
  - Boehringer Ingelheim Investigational Site 2, Trebišov
  - Boehringer Ingelheim Investigational Site, Trnava
  - Boehringer Ingelheim Investigational Site, Trstená
  - Boehringer Ingelheim Investigational Site, Vranov nad Topľou
  - Boehringer Ingelheim Investigational Site 1, Žilina
  - Boehringer Ingelheim Investigational Site 2, Žilina
- Slovenia (10):
  - Boehringer ingelheim Investigational Site 1, Ljubljana
  - Boehringer ingelheim Investigational Site 2, Ljubljana
  - Boehringer ingelheim Investigational Site 3, Ljubljana
  - Boehringer ingelheim Investigational Site 4, Ljubljana
  - Boehringer ingelheim Investigational Site 5, Ljubljana
  - Boehringer ingelheim Investigational Site 1, Maribor
  - Boehringer ingelheim Investigational Site 2, Maribor
  - Boehringer ingelheim Investigational Site 3, Maribor
  - Boehringer ingelheim Investigational Site 4, Maribor
  - Boehringer ingelheim Investigational Site 1, Šempeter pri Gorici

RESULTS

PARTICIPANT FLOW:
Groups:
- Mirapexin® (Pramipexole): The dose of Mirapexin® was selected by the neurologist upon his/her clinical judgement based on individual patient need and on recommendations given in the Mirapexin® Summary of Product Characteristics.
  mode of administration (admin.): Tablets for oral use
Period: Overall Study
Arm/Group | Mirapexin® (Pramipexole)
Started | 2448
Completed | 2335
Not Completed | 113
Not completed — Lack of Efficacy | 36
Not completed — Insufficient tolerability (IT) | 17
Not completed — Withdrawal by Subject | 18
Not completed — Other | 32
Not completed — Lack of efficacy and patient wish | 1
Not completed — IT and patient wish | 8
Not completed — Patients wish and other reason | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS)
Groups:
- Mirapexin® (Pramipexole): The dose of Mirapexin® was selected by the neurologist upon his/her clinical judgement based on individual patient need and on recommendations given in the Mirapexin® Summary of Product Characteristics. mode of admin.: Tablets for oral use.
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 2448
Age, Continuous [Mean (Full Range); unit: years] | 67.23 [31 to 97]
Sex/Gender, Customized [Number; unit: participants]
  Female | 1145
  Male | 1274
  missing | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of De-novo Patients in Whom Monotherapy With Mirapexin® Could be Successfully Initiated
Description: Successful initiation was defined as a clinical assessment of efficacy by the neurologist rated at least as "good" on a 4 point scale after 4-8 weeks Mirapexin® treatment, where:1 = very good; 2 = good; 3 = moderate; and 4 = poor.
  De-novo patients were identified by:
  those who were referred: - if 'Reason for Referral' = 'initiation of therapy' or for 'diagnostic reason' and for those not referred: - if initial pharmacotherapy = 'Mirapexin® monotherapy' (i.e., no other anti Parkinson Disease (PD) therapy)
Time Frame: 4 - 8 weeks
Population: Full Analysis set (FAS) of De-novo patients in whom monotherapy with Mirapexin® could be successfully initiated
Measure: Number; unit: Participants
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 833
Participants
  Very good | 403
  Good | 323
  Moderate | 73
  Poor | 15
  Global Clinical Assessment (GCA) missing | 19

2. Secondary Outcome: Change From Baseline in UPDRS (Unified Parkinson's Disease Rating Scale) Part I
Description: Change in UPDRS Part I score from baseline to final visit. The score ranging from 0-16 (0= no disability, 16= maximum disability)
Time Frame: Baseline and 4 to 8 weeks
Population: Full Analysis set (FAS)
Measure: Number; unit: Unit on a scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 2370
Unit on a scale | -1.20

3. Secondary Outcome: Change From Baseline in UPDRS Part III
Description: Change in UPDRS Part III score from baseline to final visit. Score ranging from 0 - 108 (0= no disability, 108 = worst disability).
Time Frame: Baseline and 4 - 8 weeks
Population: Full Analysis set (FAS)
Measure: Number; unit: Unit on a scale
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 2370
Unit on a scale | -11.18

4. Secondary Outcome: Global Clinical Assessments of Efficacy of Mirapexin® for All Patients
Description: Successful initiation was defined as a clinical assessment of efficacy by the neurologist rated at least as "good" on a 4 point scale after 4-8 weeks Mirapexin® treatment, where:1 = very good; 2 = good; 3 = moderate; and 4 = poor.
Time Frame: 4 - 8 weeks
Population: Treated set (TS)
Measure: Number; unit: Number of Participants
Arm/Group | Mirapexin® (Pramipexole)
Number analyzed (Participants) | 2448
Number of Participants
  Very good | 1043
  Good | 1004
  Moderate | 263
  Poor | 55
  Global Clinical Assessment (GCA) missing | 83

ADVERSE EVENTS:
Time Frame: During 4 - 8 weeks of therapy
Arm/Group | Mirapexin® (Pramipexole)
Serious Adverse Events (participants affected / at risk) | 0/2448
Other Adverse Events (participants affected / at risk) | 0/2448

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.